CLINICAL TRIAL: NCT04395430
Title: Adapting the US-based Clinic-community Model of Child Obesity Treatment Into an Online Intervention Model in Singapore During COVID-19
Brief Title: A Novel School-clinic-community Online Model of Child Obesity Treatment in Singapore During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke University (Other); Duke-NUS Graduate Medical School (Other); Sport Singapore (Unknown); Health Promotion Board, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190049
Record Dates: First submitted 2020-02-03; First posted 2020-05-20 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Obesity; Clinical Trial
Keywords: Exercise; Child Health; Child, Preschool; Body Mass Index; Healthy Lifestyle; Community Networks; internet-based intervention
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information Group (Active Comparator): Subjects randomized to the Information Group will receive standard care and age appropriate reading books.
  Interventions: Behavioral: Usual Care
- Intervention Group (Experimental): Subjects randomized to the Intervention Group will receive standard care plus invitation to participate in the online KKH Sports Singapore programme.
  Interventions: Behavioral: Usual Care; Behavioral: online KKH Sports Singapore Program with Usual Care

INTERVENTIONS:
Behavioral: Usual Care — Participants will receive standard care which consist of the following:
  * a lifestyle counseling visit
  * educational materials
  * goal-setting by a healthcare professional, and
  * information about general weight management resources.
  * weighing scale and measuring tape with instructions to use
  * fitness tracker
Behavioral: online KKH Sports Singapore Program with Usual Care — Participants will receive standard care and basic sports equipment and cooking materials for the online programme.
  The online programme will be available up to 4 days per week (Weekdays evenings and Weekends mornings or early afternoons) and all household family members are invited to participate. The majority of the programming will be run by trained research coordinator and volunteers from KKH and Sports Singapore coaches. A regular rotation of comprehensive programming is provided, which includes online fitness, cooking, nutrition, and peer support classes. Every session includes up to 60 minutes of exercise and/or active play, and each session has an additional special 'theme.' For example, one to two sessions per week includes nutrition related programming (e.g., cooking classes), parent specific activities (e.g., a yoga class), peer support sessions (e.g., small group discussions around issues such as weight stigmatization), and fitness classes (e.g., soccer classes).
  Arms: Intervention Group

SUMMARY:
Background: The Coronavirus 2019 (COVID-19) is an infectious disease, which was first identified in December 2019 and has then spread rapidly around the world. COVID-19 spreads mainly through respiratory droplets and causes people to experience mild to moderate respiratory illness. On 11 March 2020, the World Health Organisation (WHO) declared COVID-19 a pandemic. With the surge in cases and to contain the spread of this disease, Singapore implemented a circuit breaker to reduce movements and interactions in public and private places. People are advised to stay at home and practise social distancing. With restrictions in movements, parents and children are likely to be more sedentary in this pandemic. There is an urgent need to move face-to-face interventions to online interventions as it is important to be active in this period.

Childhood obesity threatens the health of US and Singapore populations. In the US, 30% of children are overweight, 17% have obesity, and 8% have severe obesity. In Singapore, 13% of children have obesity, and approximately half of all overweight children live in Asia. In both countries the prevalence is increasing, especially amongst the lower income populations, and is associated with future cardiovascular and metabolic disease. In US, obesity is most prevalent in Black and Hispanic populations and in Singapore, obesity affects Malays and Indians disproportionately. The underlying drivers and potential solutions thus share many common factors. The current evidence shows a clear dose-response effect with increasing number of hours of treatment, with a threshold for effectiveness at > 25 hours over a 6-month period. A key gap in delivering this recommendation is meeting the intensity, and delivering comprehensive treatment that is culturally relevant, engaging to families, and integrated within the community context.

The study is an online pilot randomised controlled trial among children aged 4-7 with obesity, in Singapore, to test a novel school-clinic-community online intervention, the KK Hospital (KKH) Sports Singapore program, for child obesity treatment with usual care. The primary outcome is intensity of treatment as measured by hours of exposure to intervention.

The online KKH Sports Singapore program involves 4-6 weekly online sessions of physical activity and nutrition lessons for children and parents.

DETAILED DESCRIPTION:
Through this trial, the investigators will address the following aims:

1. To demonstrate implementation feasibility and fidelity of the Duke community-based intervention model into an online model. The investigators hypothesise that the evidence-based implementation strategy tested in the US with Parks and Recreation will be adaptable for use at Duke-National University Singapore (NUS) with Singapore Sport, leading to online implementation within a 3-month period, and children in the intervention will receive up to 60 minutes of moderate-to-vigorous physical activity per session.
2. To meet current recommendations for intensity of obesity treatment. As compared with usual care, the investigators hypothesise that children in the online intervention will be more likely to receive >25 hours over 6 months of treatment.
3. To estimate the effectiveness of the online intervention. Children who participate in the online intervention, as compared with usual care, will demonstrate improvements in health outcomes at 6-months, including cardiorespiratory fitness, weight-related quality of life and stabilisation or reduction in BMI at 6 months.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the inclusion criteria to participate in this study.

* Overweight as defined by BMI percentile of above 90th percentile
* Age 4-7 years old in the year of referral
* Ability to provide informed consent

Exclusion Criteria:

* Patients with secondary causes of obesity especially genetic syndromes e.g. Trisomy 21, Prader-Willi
* Currently participating in a weight management program
* Unable to understand and speak English sufficiently to give informed consent and complete the research assessments.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Intensity of intervention | 6 months
  Measure intensity of intervention from baseline to 6 months. Intensity is measured using the number of hours of exposure to intervention.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline, 3 months and 6 months
  Measure change in cardiorespiratory fitness at baseline, 3 months and 6 months using the 3 minute step test.
Change in quality of life | Baseline, 3 months and 6 months
  Measure change in quality of life at baseline, 3 months and 6 months using the Paediatric Quality of Life Inventory (PedsQL; US version 4). PedsQL is a comprehensive and multi-dimensional construct that includes physical, emotional, and social functioning to assess quality of life in the children. It uses a 5-point Likert scale where 0= never, 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always. Items will be reverse scored and linearly transformed to a 0-100 scale so that higher scores indicate better quality of life.
Change in BMI | Baseline, 3 months and 6 months
  Measure the stabilisation or change in BMI at baseline, 3 months and 6 months. Body mass index (BMI) will be calculated as kg/m2.
Change in self-esteem | Baseline, 3 months and 6 months
  Measure change in self-esteem at baseline, 3 months and 6 months. Self-esteem is measured using the Behavioural Rating Scale of Presented Self-Esteem questionnaire. The first category of items consists of active displays of confidence, curiosity, initiative, exploration and independence while the second category consists of adaptive reactions to change or stress. It uses a four-point scale from 1-4 where higher scores indicate higher self-esteem.
Change in eating behaviour | Baseline, 3 months and 6 months
  Measure change in eating behaviour at baseline, 3 months and 6 months. Eating behaviour is measured using the Child Eating Behaviour Questionnaire (CEBQ). The questionnaire consists of 35 items and measures food responsiveness, emotional over-eating, enjoyment of food, desire to drink, satiety responsiveness, slowness in eating, emotional under-eating and food fussiness using a 5-point Likert scale (1= never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always). Higher scores indicate higher level of behaviour in the respective dimensions.
Change in gross motor skills | Baseline, 3 months and 6 months
  Measure change in gross motor skills at baseline, 3 months and 6 months. Gross motor skills is measured using the Test of Gross Motor Development (Ver. 3.0). The first subtest, Locomotor, measures the gross motor skills that require fluid coordinated movements of the body as the child moves in one direction or another. The second subtest, Ball Skills, measure the gross motor skills that demonstrate efficient throwing, striking, and catching movements.
Change in caloric intake | Baseline, 3 months and 6 months
  Measure change in caloric intake using a three day food diary at baseline, 3 months and 6 months.
Change in physical activity | Baseline, 3 months and 6 months
  Measure change in physical activity using results from accelerometer to assess time spent on sedentary and moderate to vigorous physical activity at baseline, 3 months and 6 months.
Change in blood pressure | Baseline, 3 months and 6 months
  Measure change in blood pressure at baseline, 3 months and 6 months. Blood pressure will be measured in mmHg via an electronic sphygmomanometer. Both systolic and diastolic blood pressure will be measured.
Change in waist circumference | Baseline, 3 months and 6 months
  Measure change in waist circumference at baseline, 3 months and 6 months. Waist circumference is measured at the narrowest point between the lower costal (rib) border and the iliac crest using a non-extensible steel tape.
Change in servings of fruits and vegetables | Baseline, 3 months and 6 months
  Measure change in number of servings of fruits and vegetables using a three day food diary at baseline, 3 months and 6 months .

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chu Shan Chew, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore